CLINICAL TRIAL: NCT02410122
Title: The Natural History of the Progression of Atrophy Secondary to Stargardt Disease Type 4 (STGD4): A Prospective Longitudinal Observational Study of Stargardt Disease Type 4, a PROM1- Related Macular Dystrophy
Brief Title: The Natural History of the Progression of Atrophy Secondary to Stargardt Disease Type 4: PROM1-Related Macular Dystrophy
Acronym: ProgStar-4
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: The Shulsky Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: NA_00092688
Record Dates: First submitted 2015-03-05; First posted 2015-04-07 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Stargardt Disease
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
While a fair amount of clinical data on Stargardt disease type 1 (STGD1) have been published, very little is known about Stargardt disease type 4 (STGD4). The ProgStar 04 study is an important opportunity to leverage the infrastructure, clinical trials sites, methods, and central reading center of the ProgStar program to investigate the progression of STGD4 and will help to establish patient cohorts worldwide for future clinical trials.

DETAILED DESCRIPTION:
The PROM1 gene codes a protein called Prominin 1 (PROM1; also known as CD133 and AC133), most known for its original use as a human stem cell-specific marker. In the retina, PROM1 is involved in the formation and organization of disks within the outer segment (OS) of the photoreceptors. It is within this particular region that most of the electrochemical signals in response to light are generated (visual cycle-phototransduction). In STGD4, mutations in the PROM1 gene result in a defective isoform of the PROM1 protein that becomes trapped in the myoid region of the photoreceptors and cannot migrate to the OS site where disks are formed. Ultimately, the absence of PROM1 in the OS affects the growth and organization of the disks, which leads to disk malfunction and to vision problems.

Although many advances in genetic science have helped to recognize this variant of STGD, a comprehensive description of the natural history, including the variability in cone and rod dysfunction, of this STGD variant is not available. While there is no known treatment for STGD at this time, the preparation for future therapeutic approaches and for planning clinical trials must include an understanding of the disease itself, its variability, its progression and its correlation with visual loss. Moreover, clinical trials that aim to slow down the progression and/or to restore vision require validated outcome measures to prove treatment efficacy. However, such outcomes have not been established for STGD overall.

In summary, the characterization of STGD4-specific clinical manifestations, progression and prognosis as well as identification of outcome measures for clinical trials are critical to develop new clinical trials for STGD4. Hence, ProgStar 4 is developed as a prospective longitudinal observational study of patients with mutations in the PROM1 gene and a phenotype consistent with STGD.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed informed consent form and authorization allowing the disclosure and use of protected health information.
2. The designated primary study eye must have at least one well-demarcated area of atrophy. The lesion size should not exceed the area to be tracked in the OCT mode (20x20 degrees).
3. Have at least one pathogenic mutation confirmed in the PROM1 gene and a Stargardt phenotype.
4. The primary study eye must have clear ocular media and adequate pupillary dilation to permit good quality FAF and sd-OCT imaging in the opinion of the investigator.
5. Be able to cooperate in performing the examinations.
6. Be willing to undergo ocular examinations once every 6 months for up to 24 months.
7. Be at least six years old.
8. Both eyes can be included if inclusion criteria are fulfilled for both eyes.

Exclusion Criteria:

1. Ocular disease, such as choroidal neovascularization, glaucoma and diabetic retinopathy, in either eye that may confound assessment of the retina morphologically and functionally.
2. Intraocular surgery in the primary study eye within 90 days prior to baseline visit.
3. Current or previous participation in an interventional study to treat STGD such as gene therapy or stem cell therapy. Current participation in a drug trial or previous participation in a drug trial within six months before enrollment. The use of oral supplements of vitamins and minerals are permitted although the current use of Vitamin A supplementation shall be documented.
4. The site Principal Investigator may declare any patient at their site ineligible to participate in the study for a sound medical reason prior to the patient's enrollment into the study.
5. Any systemic disease with a limited survival prognosis (e.g. cancer, severe/unstable cardiovascular disease).
6. Any condition that would make adherence to the examination interfere with the patient attending their regular follow-up visits schedule of once every 6 months for up to 24 months difficult or unlikely, e.g. personality disorder, use of major tranquilizers such as Haldol or Phenothiazine, chronic alcoholism, Alzheimer's Disease or drug abuse.
7. Evidence of significant uncontrolled concomitant diseases such as cardiovascular, neurological, pulmonary, renal, hepatic, endocrine or gastro-intestinal disorders.
8. Patient is known to have one or more pathogenic mutation(s) in the ABCA4, RDS, or ELOVL4 genes.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study shall enroll participants with PROM1 mutations and associated STGD4 phenotype at up to 10 clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Growth of atrophic lesions as measured by fundus autofluorescence (FAF) imaging | 24 months

SECONDARY OUTCOMES:
Growth of atrophic lesions as measured by fundus autofluorescence (FAF) imaging | 12 months
Rate of retinal thinning and photoreceptor loss as measured by spectral domain optical coherence tomography (sd-OCT) | 12 months
Rate of retinal thinning and photoreceptor loss as measured by spectral domain optical coherence tomography (sd-OCT) | 24 months
Loss of retinal sensitivity as measured by microperimetry | 12 months
Loss of retinal sensitivity as measured by microperimetry | 24 months
Change in best-corrected visual acuity by using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol | 12 months
Change in best-corrected visual acuity by using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol | 24 months
Correlation of all outcome measures with genetic profile | 12 months
Correlation of all outcome measures with genetic profile | 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Wilmer Eye Institute, Baltimore, Maryland
  - Retina Foundation of the Southwest, Dallas, Texas
- Germany (2):
  - Universitäts-Augenklinik Bonn, Bonn
  - Center for Opthalmic Research, University of Tuebingen, Tübingen
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: the Natural History of the Progression of Atrophy Secondary to Stargardt Disease (ProgStar) — http://progstar.org/progstar-home/progstar-4/